CLINICAL TRIAL: NCT03141840
Title: Clinical Trial of Safety and Efficacy of Topical ABL01 Treatment of Onychomycosis
Brief Title: Clinical Trial of Topical ABL01 Treatment of Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbell AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB001
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Onychomycosis of Toenail

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trail comparing ABL01 and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects are randomly assigned to treatment or placebo groups by a predetermined algoritm using sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Experimental group: ABL01 is to be applied topically to the infected nail once a week during the study period to counter onychomycosis.
  Interventions: Device: ABL01
- Control (Placebo Comparator): Control group: Placebo solution to be applied topically to the infected nail once a week during the study period to counter onychomycosis.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: ABL01 — Experimental medical device
  Arms: Experimental
Device: Placebo — ABL01 lacking active component
  Arms: Control

SUMMARY:
This clinical trial seeks to investigate if an experimental medical device, ABL01, can be used to treat onychomycosis. In a 1-year trial the effectiveness of ABL01 will be tested against placebo in 70 study subjects with onychomycosis of the big toe nail. The endpoint of the trial is clinical improvement and cure at the 6 and 12 month time-point.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to determine the safety and effectiveness of the medical device ABL01. The intended use of ABL01 is to reduce and treat onychomycosis, fungal nail infection. ABL01 is a solution intended to be topically administered weekly to infected nails. The trial is designed as a double blinded randomized placebo controlled clinical trial. The trial involves 70 study subjects, half of which will receive ABL01 and the other half placebo. The inclusion criteria for study subjects are adult men and women that present with distal lateral subungual onychomycosis (DSU) on the big toe nails. Furthermore, the extent of DSU should not involve more than half of the area of the nail.

The study subjects will themselves apply the study solution weekly to the treated nail. The trial will run for 6 months with a possible extension to maximum 12 months. There will be a total of 4 study visits at baseline, 3, 6 and 12 months to follow up the progress of the trial. The primary objective of the trial is to determine if ABL01 treatment are able to reduce and treat onychomycosis. Secondary objectives are to collect safety data, determine if the ABL01 are perceived as easy to use and assess long term effects of the treatment. The endpoint of the trial is reduction in clinical signs or complete cure of onychomycosis at the 6- or 12-month time-point.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Men and women above age 18 weighing over 40 kg
* Present with distal lateral subungual onychomycosis of any of the big toe nails
* The onychomycosis should involve less than 50 % of the nail bed and may not have reached the cuticle

Exclusion Criteria:

* Unable to come for study visits
* Known allergy to any of the components in ABL01
* Not willing to participate in the trial or not able to understand the content of the trial
* Present with proximal subungual onychomycosis or superficial onychomycosis.
* Present with distal lateral subungual onychomycosis of other nails than the big toe.
* More than 50 % of the nailbed affected by onychomycosis or the cuticles infected
* Known conditions (like psoriasis) that cause abnormal nail appearance
* Nail damage caused by trauma, pressure or other mechanical reasons
* Currently on immunosuppressive therapy
* Showing signs of poor peripheral blood circulation
* Used another topical antifungal treatment within 1 month of screening
* Used a systemic antifungal treatment within 3 months of screening
* Participated in any other clinical onychomycosis trial in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Number of study subjects with a reduction in infected nail area at 6 months. | 6 months
  Clinical improvement of the condition is assessed by analyzing changes in infected nail area (in relation to total nail area) due to ABL01 or placebo treatment. Clinical improvement is considered to be a 40% reduction in infected area at the 6 month time period.

SECONDARY OUTCOMES:
Questionnaire regarding subjects opinion of the treatment, nail improvement. | 12 months
  Subjects score (1-5) the perceived improvement of their nail condition.
Questionnaire regarding subjects opinion of the treatment, ease of use. | 12 months
  Subjects score (1-5) the perceived ease of using ABL01.
Number of study subjects with treatment-related adverse events | 12 months
  Subject reported safety data in combination with reported adverse events and adverse device effects related to the topical administration of ABL01.
Number of study subjects with a reduction in infected area of the nail | 12 months
  Clinical improvement of the condition is assessed by analyzing changes in infected nail area (in relation to total nail area) due to ABL01 or placebo treatment. Clinical improvement is considered to be a 80% reduction in infected area at the 12 month time period.
Number of study subjects with clinical cure | 12 months
  Clinical cure is established with a negative test for dermatophytes as assessed by DNA-analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Irini Mouratidou-Kontorinis, Principal Investigator — Fotcompaniet Stockholm
Locations (1):
- Fotcompaniet Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No